CLINICAL TRIAL: NCT06202950
Title: The Effect of Mindfulness and Yoga on Stress Level, Quality of Life and Glycemic Control in Youth With Type 1 Diabetes
Brief Title: Type 1 Diabetes,Mindfulness,Yoga,Stress,Health Quality,Glycemic İndex
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, EMİNE SARIKAMIŞ KALE, Clinical asistant, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/70
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Diabetes; Stress
Keywords: Mindfulness; Yoga; Type 1 Diabetes; Youth; Stress Level; Quality of Life; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Yoga; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga (Experimental): Applying yoga for one hour a week for eight weeks to with type 1 diabetes
  Interventions: Behavioral: Yoga
- Mindfulness (Active Comparator): Applying mindfulness to youth with type 1 diabetes one hour a week for eight weeks
  Interventions: Behavioral: Mindfulness
- control (No Intervention): the control group received the usual care

INTERVENTIONS:
Behavioral: Yoga — Applying yoga for one hour a week for eight weeks to an adolescent with type 1 diabetes
  Arms: Yoga
Behavioral: Mindfulness — Applying mindfulness for one hour a week for eight weeks to an adolescent with type 1 diabetes
  Arms: Mindfulness

SUMMARY:
The study will examine the effects of Mindfulness-Based Stress Reduction Program and yoga on stress level, quality of life and glycemic control in Youth with Type 1 diabetes.

DETAILED DESCRIPTION:
Chronic disease; It is defined as a condition that causes permanent disability, is irreversible, occurs as a result of pathological changes, requires special training, long-term care, supervision and control for the rehabilitation of the patient, and limits daily functions. According to the World Health Organization (WHO) data on chronic diseases; Every year, 41 million people in the world die due to chronic diseases, and it is stated that these numbers correspond to 74% of the deaths in the world. Nowadays, chronic diseases are becoming an increasing health problem, especially for children and adolescents. According to WHO, the incidence of chronic diseases in adolescence is reported to be 15%. According to the report published by the American Academy of Pediatrics (APA), 10-20 million children and adolescents in the United States (USA) have some kind of chronic disease.Diabetes is one of the most common non-communicable chronic diseases globally. Diabetes Mellitus (DM) is a chronic metabolic disease that develops as a result of insufficiency, deficiency and/or absence of the insulin hormone secreted from beta cells in the pancreas, is characterized by hyperglycemia, and causes disorders in carbohydrate, fat and protein metabolism. It has a chronic course and is the most common metabolic disease in childhood. Although there are different types of diabetes, Type 1 diabetes is common in childhood. Type 1 diabetes cases constitute 10-15% of all diabetic patients, and this rate is increasing. Genetic, environmental and autoimmune factors play an important role in the development of Type 1 diabetes . The incidence of the disease, which is often seen between the ages of 7-15, increases between the ages of 4-6 and 10-14. According to the 10th Diabetes Atlas data published by the International Diabetes Federation in 2021; There are 536.6 million people with diabetes worldwide, and this number is expected to increase to 783.2 million in 2045. It is reported that the number of individuals with diabetes among children and adolescents between the ages of 0-19 worldwide is approximately 1.99 million, and 1.2 million of this number consists of children and adolescents with Type 1 diabetes. In our country, it is reported that the number of children and adolescents with Type 1 diabetes between the ages of 0-18 is approximately 17 thousand and the number of adolescents with diabetes between the ages of 10-18 is approximately 13 thousand.The fact that diabetes is a disease that is not easy to manage, combined with problems such as estrangement from parents in adolescence, increased sense of independence, physiological change and peer pressure, can cause many difficulties for the adolescent in fulfilling his developmental tasks.

In studies conducted with adolescents with type 1 diabetes; In the study to determine the quality of life of healthy children/adolescents with Type 1 diabetes aged 4-15, it was found that the quality of life of children and adolescents with Type 1 diabetes was lower than that of healthy children and adolescents.

In order to determine the time management skills of adolescents with Type 1 diabetes and the effect of these skills on metabolic control, another study with 69 adolescents with Type 1 diabetes between the ages of 13-19, using the Diabetes Adolescent Diagnosis Form, Diabetes Time Management Questionnaire (DBYA), Habits and Behaviors in Adaptation to Diabetes. In the research conducted using the and Information Survey (DUADBA), Metabolic Control and Daily Record Form; It has been stated that adolescents with good time management manage diabetes better and that managing diabetes well does not affect metabolic control.study applied the Psychological Symptom Screening Test (SCL-90-R) to 56 individuals with Type 1 diabetes between the ages of 7 and 21 in order to determine the psychological symptoms and findings of children and adolescents attending a diabetes camp. As a result of this research, "50.9% of the patients had somatization, 47.3% had anxiety, 43.9% had obsession, 33.3% had depression, 37.5% had psychosis, 48.2% had It was determined that there were multiple psychiatric findings, including anger in 100% of patients and phobia in 28.1%.In the study to examine the self-concept of children/adolescents with Type 1 diabetes and their ways of coping with stress; It has been stated that self-concept is higher in those with a short duration of diabetes or 11-15 years than in those with a diabetes duration of 6-10 years, and that coping with stress was found to be higher in adolescents aged 14-17 without Type 1 diabetes than in adolescents with diabetes .

In the research conducted with 349 adolescents with Type 1 diabetes and 409 healthy individuals between the ages of 6-18 from Kuwait, in order to examine the social and psychological conditions of children/adolescents; Depression and anxiety levels of children and adolescents with type 1 diabetes were found to be higher and their psychosocial relationships were worse.In a study to examine the symptoms of depression in adolescents with Type 1 diabetes, including 45 male and 72 female adolescents with Type 1 diabetes, depressive symptoms were found in 50% of the adolescents. It has also been reported that adolescents between the ages of 14 and 16 have more depressive symptoms than younger ones.

In the study which the coping skills with anxiety and glycemic control were investigated in adolescents with Type 1 diabetes, 145 individuals were studied and the Coping Inventory of Stressful Situations was applied. In this study, it was found that as the duration of the disease increases, anxiety decreases and the ability to cope with the disease increase.In the study on the prevalence of depression and anxiety in individuals with Type 1 diabetes, the Hospital Anxiety and Depression Scale was used. In a study conducted with a total of 502 individuals, it was found that anxiety was more common than depression in individuals with Type 1 diabetes, and depression and anxiety were more common in women than in men .

In the study investigating depressive symptoms in children and adolescents with Type 1 diabetes, the Children's Depression Inventory was administered to 145 children and adolescents with Type 1 Diabetes. As a result of the research, high rates of depression were found in 15% of children and adolescents. It has also been reported that depression increases in girls and with increasing age .

In the meta-analysis study , it was stated that only 51% of patients with Type 2 diabetes reached the hemoglobin A1c (HbA1c) target of <7%. Studies on HbA1c in adolescents with type 1 diabetes are limited in number; In the HbA1c study conducted by with 66 071 children and adolescents in 8 high-income countries, it was stated that the HbA1c value varied between 7.6% and 8.8% and that HbA1c increased significantly during the transition from childhood to adolescence Type 1 diabetes; In addition to being a metabolic, chronic and organic disease, it is also a disease that has a psychosocial dimension. Studies have shown that the rate of psychiatric disorders in adults with diabetes varies between 33% and 42% and is 2-3 times higher than the general prevalence rate in society, and another study has shown that in children aged 8-17, children and adolescents with insulin-dependent Type 1 diabetes, It is stated that they have more mental difficulties than their healthy peers.Adolescents with type 1 diabetes experience physical, emotional and social problems. It is suggested that the reason for this is that both the blood sugar level and its irregularities directly affect the brain and psychological functions, and the blood sugar level is affected by psychological and emotional changes. A child/adolescent with type 1 diabetes is obliged to carry out interventions such as measuring blood sugar more than once a day, adjusting the insulin dose and administering insulin for the management of the disease, and must cope with this situation. Due to all these reasons, in adolescents with Type 1 diabetes; Depression, anxiety disorder, decrease in quality of life, eating disorder, fear of hypoglycemia, difficulty in coping and adjustment disorder may develop. Positive results are achieved with the Mindfulness-Based Stress Reduction Program and yoga practice, which are mind and body-based interventions in the process of coping with the psychosocial and physiological problems experienced by adolescents with type 1 ..diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Youth with Type 1 diabetes between the ages of 13 and 18 with a diabetes age of at least 12 months
* Not having participated in a Mindfulness-Based Stress Reduction Program or doing yoga before,
* Speaking and understanding Turkish,
* Able to read and write,
* Having no other physiological or psychological diseases,
* No mental disability,
* Not using psychoactive drugs,
* Parents volunteered for their child to participate in the research and signed the consent form,
* During the application phase, you should have eaten 1.5-2 hours before the application and your blood sugar should be between 150-200mg/dl before the application

Exclusion Criteria:

* Failed to complete the program
* Youth diagnosed with acute or chronic diseases in addition to diabetes during the study

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
10-item version of the Diabetes Stress Questionnaire for Youths with Type 1 Diabetes | 8 weeks
  use the scale with patients 12 and up and we administer it via online survey (Qualtrics). Scores vary from 0 (not at all) to 3 (very much), so the min score=0, and the max score=30. We use the clinical cut off of 12 (scores >=12 are flagged).
pediatrics quality of life inventoryTM (PedsQL) diabetes module 3.0 for Turkish adolescents with type 1 diabetes scale | 8 weeks
  The 28-item multidimensional PedsQLTM 3.0 Diabetes Module included five subscales, which are diabetes symptoms (11 items), treatment barriers (4 items), treatment adherence (7 items), worry (3 items), and communication (3 items). The format
Glycemic control form | 12 weeks
  it is an assessment tool developed to evaulate the hemoglobin A1C

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Emine Sarıkamış Kale, Batman, Merkez
  - Hasan Kalyoncu University, Gaziantep, Sahinbey

IPD SHARING:
Plan to Share IPD: Yes